CLINICAL TRIAL: NCT07223190
Title: A Phase 3, Open-label, Randomized, Controlled Trial of Subcutaneous Versus Intravenous Blinatumomab in Newly Diagnosed Adults With Philadelphia Chromosome Negative B-cell Precursor Acute Lymphoblastic Leukaemia
Brief Title: A Study Evaluating Subcutaneous Versus Intravenous Blinatumomab in Newly Diagnosed Adults With B-cell Precursor Acute Lymphoblastic Leukaemia
Acronym: AUDAX
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240113; 2025-523291-23 (EudraCT Number)
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Philadelphia Chromosome Negative B-cell Precursor Acute Lymphoblastic Leukemia
Keywords: Blinatumomab; Lymphoblastic Leukemia; HyperCVAD
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab; CVAD protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HyperCVAD + cIV Blinatumomab in Consolidation (Active Comparator): Participants with Ph-negative B-ALL will receive cIV blinatumomab infusion for cycles 1, 2, 5 and 6 (each cycle will be 35 days), in conjunction with chemotherapy (HyperCVAD) for cycles 3, 4, 7 and 8 (each cycle will be 2-4 weeks).
  Interventions: Drug: Blinatumomab; Drug: HyperCVAD
- HyperCVAD + SC Blinatumomab in Consolidation (Experimental): Participants with Ph-negative B-ALL will receive SC injections of blinatumomab for cycles 1, 2, 5 and 6 (each cycle will be 35 days), in conjunction with chemotherapy (HyperCVAD) for cycles 3, 4, 7 and 8 (each cycle will be 2-4 weeks).
  Interventions: Drug: Blinatumomab; Drug: HyperCVAD

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab will be administered as a SC injection.
  Arms: HyperCVAD + SC Blinatumomab in Consolidation
Drug: Blinatumomab — Blinatumomab will be administered as a cIV infusion.
  Arms: HyperCVAD + cIV Blinatumomab in Consolidation
Drug: HyperCVAD — HyperCVAD will administer as the chemo regimen as part of the standard of care (SOC) regimen.

SUMMARY:
The main objective of this trial is to demonstrate that subcutaneous (SC) blinatumomab in conjunction with chemotherapy (Arm B) is non-inferior to continuous intravenous infusion (cIV) blinatumomab in conjunction with chemotherapy (Arm A) in overall survival (OS) in newly diagnosed participants with Philadelphia chromosome (Ph) negative B-cell precursor acute lymphoblastic leukemia (B-ALL) who are in complete remission (CR) or CR with incomplete peripheral count recovery (CRi) after induction.

ELIGIBILITY:
Inclusion Criteria:

* Participants with newly diagnosed Philadelphia (Ph)-negative B-cell precursor acute lymphoblastic leukemia (ALL).
* Age ≥18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2, higher ECOG score allowed if due to underlying leukemia.
* Adequate organ function as described below:

  * Renal: estimated glomerular filtration rate (GFR) ≥30 mL/min/1.73m^2 per the Modification of Diet in Renal Disease for adult participants equation
  * Hepatic function: total bilirubin ≤3.0 mg/dL prior to start of treatment; unless due to Gilbert's Disease or if liver involvement with leukemia
  * Cardiac: left ventricular ejection fraction (LVEF) ≥50% and no clinically significant, uncontrolled, or active cardiovascular, cerebrovascular, or peripheral vascular disease, or history of or active venous thromboembolism (VTE) disease.

Exclusion Criteria:

Other Medical Conditions

* Isolated extramedullary disease.
* History or presence of clinically relevant central nervous system (CNS) pathology or event such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis.
* Current autoimmune disease or history of autoimmune disease with potential CNS involvement.
* History of other malignancy within the past 3 years, except for malignancy treated with curative intent with low risk for recurrence. Exceptions include:

  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated cervical carcinoma in situ without evidence of disease.
  * Adequately treated breast ductal carcinoma in situ without evidence of disease.
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer.
  * Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.
* Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B or hepatitis C virus.
* Participant with symptoms and/or clinical signs and/or radiographic and/or sonographic signs that indicate an acute or uncontrolled chronic infection, any other concurrent disease or medical condition that could be exacerbated by the treatment or would seriously complicate compliance with the protocol.

Prior/Concomitant Therapy • Prior cancer chemotherapy/immunotherapy for this newly diagnosed B-ALL before the start of protocol-required therapy with the exception of intrathecal (IT) chemotherapy or pre-phase chemotherapy. Localized radiation for pain or disease control is allowed.

Prior/Concurrent Clinical Trial Experience

•Currently receiving a trial intervention, or less than 30 days or 5 half-lives if known (whichever is later) since ending a trial intervention in another investigational device or drug trial.

Other Exclusions

* History or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator, would pose a risk to participant safety.
* Female participants of childbearing potential unwilling to use contraception.
* Female participants who are breastfeeding or who plan to breastfeed.
* Female participants planning to become pregnant or donate eggs.
* Female participants of childbearing potential with a positive pregnancy test assessed at screening by a highly sensitive urine or serum pregnancy test.
* Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception.
* Male participants with a pregnant partner who are unwilling to practice abstinence or use a condom.
* Male participants unwilling to abstain from donating sperm.
* Participant has known sensitivity to any of the products or components to be administered during dosing.
* Participant considered unlikely to be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, Clinical Outcome Assessments) to the best of the participant and investigator's knowledge; exception - unavailability of a patient-reported outcome (PRO) in the participants' preferred/native language is not prohibitive to enrollment for eligible participants.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2033-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 5 years from randomization

SECONDARY OUTCOMES:
Number of Participants who Experience Treatment-emergent Adverse Events (TEAEs) | Up to 5 years from randomization
  Number of participants who experience TEAEs, serious TEAEs, treatment-related adverse events, and adverse events of interest.
Area Under the Concentration-time Curve in Cycle 1 (AUCcycle 1) for SC Blinatumomab | Up to Cycle 1 Day 35 (Cycle length = 35 days)
AUCcycle 1 for cIV Blinatumomab | Up to Cycle 1 Day 35 (Cycle length = 35 days)
Average Concentration Following Cycle 1 Day 19 Dosing (Cavgd19dose) for SC Blinatumomab | From predose on Cycle 1 Day 19 to predose on Cycle 1 Day 22 (Cycle length = 35 days)
Steady-state Concentration (Css) for cIV Blinatumomab | Up to Cycle 1 Day 29 (Cycle length = 35 days)
Relapse-free Survival (RFS) | Up to 5 years from randomization
  RFS is defined as time from randomization until relapse, death from any cause or measurable residual disease (MRD) non-response, whichever is earlier.
Number of Participants With CR With MRD Response | Up to 5 years from randomization
  CR with MRD response is defined as MRD <10^-4. CR with MRD response is defined as <5% bone marrow (BM) blasts by cytomorphology with full recovery of peripheral blood counts (absolute neutrophil count [ANC] >1000/µl and platelets >100,000/µl) and MRD < 10^4 and no evidence of extramedullary disease (EMD).
Number of Participants With Deep CR With MRD Response | Up to 5 years from randomization
  Deep CR with MRD response is defined as MRD <10^-6. Deep CR with MRD response is defined as <5% BM blasts by cytomorphology with full recovery of peripheral blood counts (ANC > 1000/µl and platelets > 100,000/µl) and MRD ≤ 10^6 and no evidence of extramedullary disease.
Change from Day 1 Consolidation Cycle 1 to End of Consolidation in Role Functioning as Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Consolidation Cycles 1, 2, 5 and 6 Day 1 (Cycles length=35 days); Consolidation Cycles 3, 4, 7 and 8 Day 15 (Cycles length=2-4 weeks); Maintenance Cycle 1 Day 1 (Cycle length=28 days)
Change from Day 1 Consolidation Cycle 1 to End of Consolidation in Overall Quality of Life as Measured by EORTC QLQ-C30 | Consolidation Cycles 1, 2, 5 and 6 Day 1 (Cycles length=35 days); Consolidation Cycles 3, 4, 7 and 8 Day 15 (Cycles length=2-4 weeks); Maintenance Cycle 1 Day 1 (Cycle length=28 days)
Change from Day 1 Consolidation Cycle 1 to End of Consolidation in All Other Domains/Items as Measured by EORTC QLQ-C30 | Consolidation Cycles 1, 2, 5 and 6 Day 1 (Cycles length=35 days); Consolidation Cycles 3, 4, 7 and 8 Day 15 (Cycles length=2-4 weeks); Maintenance Cycle 1 Day 1 (Cycle length=28 days)
Change From Day 1 Consolidation Cycle 1 to End of Consolidation in the Visual Analogue Scale (VAS) | Consolidation Cycles 1, 2, 5 and 6 Day 1 (Cycles length=35 days); Consolidation Cycles 3, 4, 7 and 8 Day 15 (Cycles length=2-4 weeks); Maintenance Cycle 1 Day 1 (Cycle length=28 days)
  Change in the VAS will be measured from European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L).
Percentage of Time on Treatment With High Side Effect Bother From Consolidation Cycle 1 to End of Consolidation | Consolidation Cycle 1 up to Day 8 and then weekly until end of Consolidation Cycle (Cycle length = 35 days)
  Percentage of time on treatment with high side effect bother (score 3-4) from consolidation cycle 1 to end of consolidation will be measured by Functional Assessment of Chronic Illness Therapy (FACIT) GP5.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com